CLINICAL TRIAL: NCT03749915
Title: A Single Blinded Observational Study of the Effectiveness of a Pain Ease Local Anesthetic Spray, Combined With Ametop Gel, to Reduce the Discomfort of Intravenous Insertion
Brief Title: Ametop Compared to Ametop With Pain Ease Spray
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Stephan Malherbe, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H18-02364
Record Dates: First submitted 2018-11-16; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Analgesia; Topical Anesthetic
Keywords: Pain Ease; Ametop Gel
MeSH Terms: conditions — Agnosia | interventions — Tetracaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Comparator: Ametop only (Active Comparator): Ametop Gel applied as sole topical anesthetic.
  Interventions: Drug: Ametop
- Intervention: Pain Ease Cold Spray (Experimental): Pain Ease Cold spray applied immediately before IV insertion, as an adjunct to Ametop Gel.
  Interventions: Device: Pain Ease Cold Spray

INTERVENTIONS:
Device: Pain Ease Cold Spray — Pain Ease is a spray containing 1,1,1,3,3-Pentafluoropropane (HFC-245fa) and 1,1,1,2-Tetrafluoroethane (HFC-134a). It is a vapocoolant for use as a topical anesthetic.
  Arms: Intervention: Pain Ease Cold Spray
Drug: Ametop — Tetracaine Hydrochloride Gel 4%
  Other Names: Ametop Gel
  Arms: Comparator: Ametop only

SUMMARY:
The investigators propose to examine if Pain Ease spray, used as an adjunct to the topical anesthetic Ametop Gel, can improve the percentage of pain-free IV starts.

DETAILED DESCRIPTION:
Purpose:

The aim of this study is to assess the effectiveness of Pain Ease® spray, used as an adjunct to Ametop Gel™.

Hypothesis:

The investigators hypothesize that using Pain Ease® spray as an adjunct to the standard use of Ametop Gel™ will increase the number of pain free venipunctures from 30% to 50% or more.

Objectives:

Primary Objective

1. To determine if using Pain Ease® spray as an adjunct to Ametop Gel™ will increase the number of pain free venipunctures Secondary Objectives
2. To document the side effects of Pain Ease® spray and Ametop Gel™
3. To document the number of attempts for a successful IV insertion

Research Design:

The investigators propose a patient-blinded randomized control trial of Ametop Gel™ with and without Pain Ease® spray as an adjunct.

Statistical Analysis:

An interim analysis will be performed at the study's halfway point after recruitment of 120 participants. A score on the Faces Pain Scale - Revised (FPS-R) of either 0 or 2 will be considered a pain-free IV start, while a score of 4-10 will be considered a painful IV cannula insertion. Fischer's Exact test will be used to determine statistical significance; a critical alpha of 0.05 will be considered for significance.

ELIGIBILITY:
Inclusion Criteria:

* ASA I & II
* Elective day case procedure requiring an IV

Exclusion Criteria:

* Planned IV insertion after inhalation induction
* Developmental delay or inability to interpret the Revised Faces Pain Scale (FPS-R)10
* Ametop Gel™ application < 30 minutes before estimated IV start at time of screening
* Allergies to any of the components in Ametop Gel™, Pain Ease® spray, or adhesives
* Patients receiving sedative pre-medication
* Severe Needle phobia

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2018-11-20 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain-free IV insertion | intraoperative
  The number of pain free IV insertions as measured by participant indicating 0 or 2 on the Faces Pain Scale - Revised.

SECONDARY OUTCOMES:
Insertion attempts | intraoperative
  Total number of insertion attempts required for successful placement of IV cannula
FPS-R pain score | intraoperative
  Mean Faces Pain Scale - Revised pain score by group. 0-10 pain score of 0 being no pain and 10 being most pain ever experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Malherbe, FRCA, Principal Investigator — BC Children's Hospital, Department of Anesthesia
Locations (1):
- BC Children's Hospital - Department of Anesthesia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Pediatric Anesthesia Research Team website — http://part.bcchr.ca